CLINICAL TRIAL: NCT06958835
Title: Combination Antibiotic Treatment With Linezolid for Staphylococcus Aureus Bacteraemia: a Randomised Controlled Trial
Brief Title: Linezolid Plus Standard of Care
Acronym: LIPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-00655; am23Khanna3
Record Dates: First submitted 2025-04-01; First posted 2025-05-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Staphylococcus Aureus Bloodstream Infections (BSI; Bacteremia)
Keywords: Virulence factors; Linezolid; Bloodstream Infection; Hierarchical composite endpoint; Staphylococcus aureus; Bacteremia; Bacteraemia; Methicillin-resistant Staphylococcus aureus (MRSA); Penicillin-susceptible Staphylococcus aureus (PSSA); Methicillin-susceptible Staphylococcus aureus (MSSA)
MeSH Terms: conditions — Bacteremia; Sepsis; Staphylococcal Infections; Toxemia | interventions — Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linezolid (Experimental): 600mg twice a day for 5 days (in addition to the standard antibiotic treatment)
  Interventions: Drug: Linezolid 600 mg
- Placebo (Placebo Comparator): oral placebo tablets twice a day for 5 days (in addition to the standard antibiotic treatment)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linezolid 600 mg — linezolid 600 mg tablets (twice a day for 5 days)
  Arms: Linezolid
Drug: Placebo — Placebo tablets (twice a day for 5 days)
  Arms: Placebo

SUMMARY:
The aim of the study is to assess whether targeting virulence factors by administering linezolid in addition to standard antibiotic treatment improves outcomes in patients with Staphylococcus aureus bacteraemia.

DETAILED DESCRIPTION:
Staphylococcus aureus (S. aureus) is one of the deadliest bacterial pathogens, especially in high-income countries, and causes bloodstream infections (bacteraemia) in 20-30 per 100,000 people annually. Despite widely available antibiotic treatments, the 90-day mortality rate remains high at 20-30%, and complications such as organ damage, relapses, and long-term impairment affect many survivors. Existing treatments have failed to improve survival rates highlighting the urgent need for novel therapeutic strategies.

Virulence factors produced by S. aureus facilitate bacterial persistence and spread, and tissue damage. Preclinical research suggests that inhibiting the production of virulence factors may improve patient outcomes. While some clinical guidelines recommend this approach for toxin-mediated infections, randomized controlled trials (RCTs) evaluating this approach in S. aureus bacteraemia have not yet been conducted.

Linezolid, an antibiotic commonly used for pneumonia and complicated skin and soft-tissue infections, has shown strong inhibition of the expression of S. aureus virulence factors in preclinical studies. Studies in animal models demonstrated that linezolid, when combined with other antibiotics, enhances treatment efficacy and reduces bacterial toxin production. Observational studies suggest that early initiation of linezolid may lead to better patient outcomes, but no RCT has tested this approach in S. aureus bacteraemia.

This placebo-controlled trial will evaluate whether adding a 5-day course of linezolid to standard antibiotic therapy improves clinical outcomes in patients with S. aureus bacteraemia.

ELIGIBILITY:
Inclusion criteria:

* Staphylococcus aureus (S. aureus) grown from at least one blood culture
* Hospitalised at a participating centre
* ≥18 years old
* Written informed consent or fulfilling criteria for an emergency exception from informed consent requirements

Exclusion criteria:

* Administration of the initial drug treatment not feasible within 72 hours since the collection of the first positive blood culture with S. aureus
* Documented history of positive blood cultures for S. aureus occurring between 72 hours and 180 days prior to the eligibility assessment
* Necrotising fasciitis
* Currently receiving linezolid or clindamycin
* Use of any monoamine oxidase A or B inhibitor within the last two weeks
* Known hypersensitivity to linezolid or any other ingredients of the study drugs
* Current severe thrombocytopenia (i.e. <30 x 10^9/L)
* Application of study drug not possible (per mouth or per gastric tube)
* Currently breastfeeding
* Local treating team believes that death is imminent and inevitable
* Patient is receiving end of life care and antibiotic treatment is not considered appropriate
* Local treating team believes that participation in the study is not in the best interest of the patient
* Any indication that the patient is unwilling to participate in the study including an advance directive stating such unwillingness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Desirability of Outcome Ranking (DOOR) | From randomisation (day 1) until day 90
  The hierarchical composite endpoint DOOR will be calculated based on the following 4 criteria:
  1. Alive at 90 days
  2. Return to usual level of function by day 90
  3. None of the following complications: Microbiological or clinical failure leading to treatment change; Serious adverse reaction; Adverse event leading to study drug discontinuation
  4. Hospital length of stay
  The primary outcome will be expressed as the win ratio, i.e., the ratio of the number of times that participants in the intervention group have a lower DOOR compared to those in the control group.
  In this study, a pairwise comparison is used, i.e., every participant in the linezolid group is compared with every participant in the control group. When comparing two participants, the winner will be determined by the first component of the DOOR in which the two participants differ, the only exceptions being ties when both participants die or if they do not die but have the same length of hospitalisation.

SECONDARY OUTCOMES:
All-cause mortality | From randomisation (day 1) until day 90
  Proportion of patients who died from any cause during the duration of the study.
Time to death | From randomisation (day 1) until day 90
Level of function | From randomisation (day 1) until day 90
  Proportion of participants back to their usual level of function prior to the infection.
Number of participants with microbiological failure leading to treatment change | From day 14 to day 90 (randomisation = day 1)
  Any positive sterile site culture with Staphylococcus aureus (S. aureus) between 14 and 90 days after randomisation that leads to a change in treatment. A sterile site means any site of the body where microorganisms are usually absent, i.e. below the outer and inner colonised surfaces of the skin and mucous membranes. Positive sterile sites cultures include deep visceral and musculoskeletal abscesses obtained in a sterile manner.
Number of participants with early microbiological failure leading to treatment change | From day 5 to day 13 (randomisation = day 1)
  Any positive sterile site culture with S. aureus between 5 and 13 days after randomisation that leads to a change in treatment. A sterile site means any site of the body where microorganisms are usually absent, i.e. below the outer and inner colonised surfaces of the skin and mucous membranes. Positive sterile sites cultures include deep visceral and musculoskeletal abscesses obtained in a sterile manner.
Number of participants with clinical failure leading to treatment change | From day 14 to day 90 (randomisation = day 1)
  Newly identified focus of S. aureus between 14 and 90 days after randomisation as determined by the site investigator (or delegated physician) that leads to a change in treatment. This can incorporate clinical, radiological, microbiological and pathological findings.
Number of participants with early clinical failure leading to treatment change | From day 5 to day 13 (randomisation = day 1)
  Newly identified focus of S. aureus between 5 and 13 days after randomisation as determined by the site investigator (or delegated physician) that leads to a change in treatment. This can incorporate clinical, radiological, microbiological and pathological findings.
Hospital length of stay | From randomisation (day 1) until day 90
  Duration of the index acute hospital stay from randomisation until the day of hospital discharge. Transfers to another acute care hospital for continuation of acute treatment will be included in the assessment of hospital length of stay. Days after transfer to rehabilitation centres or switch to outpatient parenteral ambulatory treatment will not be included in the acute hospital stay.
Time to being discharged alive | From randomisation (day 1) until day 90
  For participants who die during the hospitalisation, 90 days will be recorded.
Days alive without being on the Intensive Care Unit (ICU) | From randomisation (day 1) until day 90
  Number of days a participant is alive and not hospitalised in the Intensive Care Unit.
Days alive without antibiotics | From randomisation (day 1) until day 90
  Number of days a participant is alive and not on any antibiotics.
Mental health | At day 90 (randomisation = day 1)
  Mental health assessed by patient-reported outcome using Short Form-36 (SF-36) questionnaire. The SF-36 questionnaire score ranges from 0 to 100, with higher scores indicating better health.
Physical health | At day 90 (randomisation = day 1)
  Physical health assessed by patient-reported outcome using SF-36 questionnaire. The SF-36 questionnaire score ranges from 0 to 100, with higher scores indicating better health.
Number of participants with persistent bacteraemia | At day 5 (randomisation = day 1)
  S. aureus-positive blood culture on day 5 (±1 day) after randomisation. If day 2 or day 3 blood cultures are negative and no subsequent blood cultures are performed, the day 5 blood culture is presumed to be negative.
Two or more systemic inflammatory response syndrome (SIRS) criteria fulfilled | At day 5 (randomisation = day 1)
  SIRS criteria:
  * Abnormal body temperature (<36°C or >38°C)
  * tachypnoea or mechanical ventilation (RR>20 breaths per minute)
  * tachycardia (HR >90 beats per minute in an adult
  * abnormal leukocyte count (from routine blood sampling on day 5 ±1 day, defined as >12.0 x 10^9/L or <4.0 x 10^9/L or >10% of immature (band) forms)
Change in C-reactive protein (CRP) | From randomisation (day 1) until day 5
  Day 1 CRP means any blood CRP measurement taken on randomisation day 1 or the calendar day prior to randomisation. If there is more than one measurement, the value recorded is the one taken closest before randomisation.
Development of new antibiotic drug resistance in Staphylococcus aureus | From randomisation (day 1) until day 90
  Any new resistance absent in the S. aureus from the initial blood culture and detected in any S. aureus cultured after the start of the intervention.
Adverse events leading to study drug discontinuation | From randomisation (day 1) until day 5
  Any adverse event (irrespective of grade) leading to study drug discontinuation as documented by the treating physician.
Serious adverse reactions until day 90 | From randomisation (day 1) until day 90
  Any serious adverse event will be reported to the study-site principal investigator, who then assesses whether there is a reasonable causal relationship with the investigational medicinal product.
Clinical signs of serotonin toxicity | From randomisation (day 1) until day 7
  Assessed using the Hunter Serotonin Toxicity Criteria.
Laboratory signs of myelosuppression | From randomisation (day 1) until day 7
  Laboratory confirmation of thrombocytopenia, anaemia, or leukopenia.
Evidence of hyperlactatemia | From randomisation (day 1) until day 7
  In case of clinical suspicion of hyperlactatemia, lactate levels will be measured and compared to specific laboratory-defined reference ranges. For increased lactate levels, the causality with the study treatment will be assessed.
Acute kidney injury | From randomisation until day 14
  Assessed on day 5 and, if participant remains hospitalised, on day 14, using the Kidney Disease Improving Global Outcomes (KDIGO) definition.
Number of participants with Clostridioides difficile (C. difficile)-associated diarrhoea | From randomisation (day 1) until day 90
  This means a stool submitted to a clinical laboratory has tested positive for C. difficile toxin or toxin gene.

OTHER OUTCOMES:
Linezolid trough plasma concentrations at day 4 or 5 | At day 5 (day of randomisation = day 1)
  Additional exploratory laboratory outcome for a subset of participants only in participating centres (results may be reported in a publication separate from the publication of the main study results).
Molecular mechanisms of S. aureus bacteraemia | From randomisation (day 1) until day 90 or until the date of the participant's first blood culture negative for S. aureus, whichever came first.
  Basic research on the location of S. aureus in human blood (extracellular or intracellular). This will be conducted in a sub-sample of participants consenting to additional blood sampling and published separately from the publication of the main study results.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kühl, PD Dr. med., Principal Investigator — University Hospital, Basel, Switzerland; Benjamin Speich, PD, PhD, Principal Investigator — University Hospital, Basel, Switzerland; Nina Khanna, Prof. Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (12):
- Switzerland (12):
  - Kantonsspital Aarau (KSA), Aarau, Canton of Aargau
  - St. Claraspital, Basel, Canton of Basel-City
  - Hôpitaux universitaires de Genève (HUG), Geneva, Canton of Geneva
  - Hôpital du Jura, Delémont, Canton of Jura
  - Centre hospitalier universitaire vaudois (CHUV), Lausanne, Canton of Vaud
  - Kantonsspital Winterthur (KSW), Winterthur, Canton of Zurich
  - Ente Ospedaliero Cantonale (EOC), Lugano, Canton Ticino
  - University Hospital Basel (USB), Basel
  - Inselspital Bern, Bern
  - HOCH Health Ostschweiz, Kantonsspital St.Gallen, Sankt Gallen
  - Stadtspital Zürich Triemli, Zurich
  - Universitätsspital Zürich (USZ), Zurich

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Study Protocol (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT06958835/Prot_001.pdf